CLINICAL TRIAL: NCT04401878
Title: Verification of Sphenopalatine Ganglion Block Success Using Transcranial Doppler in Management of Patients With Post Dural Puncture Headache
Brief Title: SGB in Management of Patients With PDPH Using TCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer, Anesthesia and Surgical Intensive Care department, Faculty of Medicine, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6140; 6140 (Other: Faculty of Medicine, Zagazig University)
Record Dates: First submitted 2020-05-18; First posted 2020-05-26 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Post-Dural Puncture Headache
Keywords: Accidental dural puncture; Post dural puncture headache; Sphenopalatine ganglion block; Transcranial Doppler
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Lidocaine; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: This study is carried out in the Orthopedic unit and included 120 patients divided into two groups: the treatment group (A) and the control group (B). Group A recruit 60 patients with a past history of epidural anesthesia who suffered from of PDPH within five days after the dural puncture. Group B included 60 patients with a history of epidural anesthesia with no PDPH.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double (Care Providor, Outcome Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment group (A) (Experimental): Patients who have PDPH are manged by SPGB, they are assessed by NRS before the block, at 30 mins, 2h, 4h, 6h, 12h, and 24hours after block. The patients are also examined by TCD before and after the block.
  Interventions: Drug: Sphenopalatine Ganglion Block using 2% lidocaine
- control group (B) (Experimental): The control group (B) of 60 patients with no PDPH were examined by TCD
  Interventions: Drug: Sphenopalatine Ganglion Block using 2% lidocaine

INTERVENTIONS:
Drug: Sphenopalatine Ganglion Block using 2% lidocaine — Sphenopalatine Ganglion Block is performed by a hollow culture swab that is connected with a 21-gauge syringe filled with three ml 2% lidocaine, inserted parallel to the floor of the nose until resistance is felt. The swab is at the posterior pharyngeal wall superior to the middle turbinate. The applicator was kept in the nostril for five to ten mins. The same procedure is done also in the second nostril. The patients are then examined by TCD.
  Other Names: Transcranial Doppler (TCD) is also utilized

SUMMARY:
This study aims to investigate the ability of SPGB in the management of PDPH. Transcranial Doppler is also used as an measure to assess the block success by detecting the variability in the cerebral hemodynamics before and after the block.

DETAILED DESCRIPTION:
This clinical trial is performed in postoperative orthopedic unit. In this study, 120 patients were enrolled who had an epidural anesthesia; 60 patients who developed PDPH joined the treatment group (A) and received the SP block. They are assessed before the procedure by NRS and at 30 mins, 2h, 4h, 6h, 12h, and 24h after the procedure. Patients are also assessed by TCD before and after the block. The control group (B) included 60 patients with no PDPH.

ELIGIBILITY:
Inclusion Criteria:

* patients are considered who had an epidural anesthesia
* Patients with ASA 1 and 2
* Patients' age ranged from 18 to 60 years.

Exclusion Criteria:

* Patients with septal perforation, nasal septum deviation,or nasal bleeding.
* Patients have recent nasal trauma
* Patients have recent nasal surgery
* Patients have a nasal infection
* Patients within ASA 3 and 4
* Patients older than sixty yrs or younger than eighteen yrs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
pain changes assessment by numeric rating scale (NRS) | Before the block and at 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours after the block
  Pain score changes are assessed before and after the block using NRS in which zero is no pain and ten is worst pain imagined. pain was assessed throughout 24 hours after performing the block and Pain relief is considered when NRS ≤ 4.

SECONDARY OUTCOMES:
Detecting the changes in cerebral vessels caliber after doing SPGB | TCD measurements are performed before SPGB is given to both groups, it is repeated again within an hour after the block for group (A) only.
  Siemens Acuson X300 ultrasound with P 4-2 phased array 2MHz probe was utilized. For all patients, both middle cerebral arteries were insonated through the transtemporal window over the zygomatic arch in front of the tragus of the ear at a depth of 50-60 mm. Tracings were also recorded for at least 10 cardiac cycles

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Abdelhaleem, MD, Principal Investigator — Faculty of Medicine, Zagazig University, Zagazig, Egypt.
Locations (1):
- Faculty of Medicine, Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
it will be available after completion of study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available 3 months after publication of study
Access Criteria: By contacting the principal investigator
URL: https://ClinicalTrials.gov

REFERENCES:
- [Background] Basurto Ona X, Osorio D, Bonfill Cosp X. Drug therapy for treating post-dural puncture headache. Cochrane Database Syst Rev. 2015 Jul 15;2015(7):CD007887. doi: 10.1002/14651858.CD007887.pub3. PMID 26176166
- [Result] Abdelhaleem NF, Othman HA, Abdel Razek GM, et al. (2019). Is the Combination of Glasgow Coma Scale and Transcranial Doppler Pulsatility Index Improving the Prediction of Outcome in Traumatic Brain Injury Patients? ZUMJ, 2019, 25(5): 529-538, doi:10.21608/zumj.2019.10082.10740